CLINICAL TRIAL: NCT02848742
Title: Evaluation of a New Dermal Cryotherapy System for the Treatment of Benign Pigmented Lesions
Brief Title: Dermal Cryotherapy for Treatment of Pigmented Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: R2 Dermatology (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2-16-001
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Pigmented Skin Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- Treatment with cryotherapy device (Experimental): To include subjects with one or more benign pigmented lesions who are willing to have the pigmented skin exposed to cooling with the Dermal Cooling System.
  Interventions: Device: Dermal Cooling System

INTERVENTIONS:
Device: Dermal Cooling System — Dermal cryotherapy

SUMMARY:
Study to evaluate the ability of the Dermal Cooling System to reduce pigmentation in benign pigmented lesions.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, multi-center study of the Dermal Cooling System to verify that the device causes a reduction in pigmentation in benign pigmented lesions, and to determine at what parameters the device is most effective.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects > 18 years of age.
2. Subject has one or more benign pigmented lesions (e.g., solar lentigines, melasma, freckles, café au lait, nevi, or hyperpigmentation), in an area suitable for treatment
3. Subject is willing to have up to 40 treatment sites and/or an area up to 8 square inches treated depending on the size and nature of the lesions identified.
4. Subject is willing to have digital photographs taken of the treatment area and agrees to use of photographs for presentation, educational, or marketing purposes.
5. Subject is willing to cover treated area or have very limited sun exposure and use an approved sunscreen of SPF 50 or higher on the treated areas for the duration of the study, including the follow-up period, if requested.
6. Subject has read and signed a written informed consent form.

Exclusion Criteria:

1. Physician prescribed medical or surgical treatment, or use of over-the-counter products to alter skin color, in the area of intended treatment in the previous 6 months (e.g., hydroquinone, corticosteroids, laser surgery)
2. Artificial tanning in the area of intended treatment within 1 month (e.g., spray, lotion, tanning bed) or intention to use artificial tanning within the follow-up period
3. Scars or tattoos in the location of the treatment sites
4. History of vitiligo, eczema, or psoriasis in the area of treatment
5. History of melanoma
6. Known history of illness or adverse reaction to cold insult (e.g., cryoglobulinemia, cold urticaria, paroxysmal cold hemoglobinuria, Reynaud's disease.
7. History of abnormal wound healing or abnormal scarring
8. Inability or unwillingness to comply with the study requirements.
9. Current enrollment in a clinical study of any other unapproved investigational drug or device.
10. Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2016-06; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Reduction of pigmentation in treated lesions | 90 days
  Changes in pigmentation graded using a 4-point standardized scale

SECONDARY OUTCOMES:
Evaluation of device- or procedure-related adverse events | 0 to 12 months
  Side effects, discomfort assessments both during treatment and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Tatsutani, PhD, Study Director — R2 Dermatology, Inc.
Locations (2):
- Diablo Clinical Research, Walnut Creek, California, United States
- Arbutus Laser Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No